CLINICAL TRIAL: NCT02023554
Title: A Pharmacokinetic Drug Interaction Study to Evaluate the Effect of Azithromycin on the Steady-State Plasma Levels of Theophylline in a Chinese Population
Brief Title: Drug Interaction Study of Azithromycin and Theophylline
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zhujiang Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 81302846-1
Record Dates: First submitted 2013-12-23; First posted 2013-12-30 (Estimated); Last update posted 2014-08-19 (Estimated); Status verified 2014-08

CONDITIONS: Chronic Obstructive Pulmonary Disease; Asthma
Keywords: azithromycin; theophylline; CYP3A4
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Asthma | interventions — Theophylline; Azithromycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Theophylline with azithromycin (Experimental): steady-state plasma concentration of theophylline in the presence of azithromycin
  Interventions: Drug: Theophylline with azithromycin
- Theophylline alone (Active Comparator): steady-state plasma concentration of theophylline alone
  Interventions: Drug: Theophylline alone

INTERVENTIONS:
Drug: Theophylline with azithromycin — Drug: Theophylline(100mg,sustained release tablets). Multi-dose of theophylline(100mg,twice daily) will administered at 8 am and 8 pm from day 1 to day 7.
  Drug:Azithromycin(250mg, capsules). Multi-dose of azithromycin(500mg,once daily) will administered at 8 pm from day 1 to day 7.
  Arms: Theophylline with azithromycin
Drug: Theophylline alone — Drug: Theophylline(100mg,sustained release tablet). Multi-dose of theophylline(100mg,twice daily) will administered at 8 am and 8 pm from day 8 to day 14.
  Arms: Theophylline alone

SUMMARY:
Macrolides are potent inhibitors of cytochrome P450 isoenzyme 3A4（CYP3A4）and thus interfere with the pharmacokinetics of many other drugs that are metabolised by this enzyme like theophylline.The aim of this study is to determine whether azithromycin can effect theophylline metabolism in patients.

DETAILED DESCRIPTION:
In this non-blinded,auto-control study,patients with Chronic Obstructive Pulmonary Disease（COPD）or asthma will serve as their own controls during the 2-week treatment phase.The subjects will be co-administered oral doses of sustained release theophylline (100mg tablets,twice daily) and azithromycin (2x250mg capsules,once daily )in the first week.Then patients will received theophylline therapy alone with the same dose in the second week.Blood samples for the measurement of theophylline plasma concentrations will be collected on Days 8 and 15 prior to dosing.All adverse events whether elicited by query, spontaneously reported or observed by clinic staff will be evaluated by the investigator and reported in the subject's case report form.

ELIGIBILITY:
Inclusion Criteria:

* patients with COPD or asthma，aged 18-75 years;
* regularly visiting our hospital;
* meeting the indications for azithromycin and theophylline simultaneously;

Exclusion Criteria:

* patients with renal or hepatic dysfunction;
* patients with congestive heart failure;
* patients with hypothyroidism or hyperthyroidism;
* patients taking drugs likely to affect the theophylline metabolism in the preceding week;
* patients with severe chronic obstructive pulmonary disease,asthma or respiratory infection;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2013-12; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
steady-state plasma concentration of theophylline | blood samples for theophylline will be collected on Days 8 and 15 before dosing
  Theophylline and it's metabolite(1,3-dimethyluric) blood concentration

CONTACTS AND LOCATIONS:
Overall Officials: Liqing Wang, Doctor, Principal Investigator — Zhujiang Hospital,Southern Medical Unversity
Locations (1):
- Zhujiang Hospital,Southern Medical Universtiy, Guangzhou, Guangdong, China